CLINICAL TRIAL: NCT01774578
Title: An Open-label, Randomized Phase IIB/III Active Control Study of Second-line Tergenpumatucel-L (Hyper-Acute(R)-Lung ) Immunotherapy Versus Docetaxel in Progressive or Relapsed Non-Small Cell Lung Cancer
Brief Title: Immunotherapy Study in Progressive or Relapsed Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG0301; 1209-1184 (Other: Office of Biotechnology Activities)
Record Dates: First submitted 2013-01-07; First posted 2013-01-24 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Non-small Cell Lung Cancer; Progression of Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Recurrent
Keywords: Non-small Cell Lung Cancer; Vaccine Therapy; Immunotherapy; Second line therapy; Progressive; Relapsed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Docetaxel; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Docetaxel (Active Comparator): Arm 1: Docetaxel 75 mg/m^2 IV given every 3 weeks x 4 doses. If response or stable: Observe until disease progression.
  First Progression: Gemcitabine 1250 mg/m^2/week for 2 weeks with 1 week rest or Pemetrexed 500 mg/m^2 every 3 weeks until disease progression or significant toxicity.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Pemetrexed
- Arm 2a: HyperAcute®-Lung Immunotherapy (weekly) (Experimental): Arm 2a: 300 Million HAL cells given by intradermal injection weekly for 11 weeks and then every 2 months for 5 additional doses.
  Up to 16 total immunizations of 300 million immunotherapy cells until disease progression or toxicity.
  First Progression: Docetaxel 75 mg/m^2 IV given every 3 weeks or Gemcitabine 1250 mg/m^2 for 2 weeks with 1 week rest or Pemetrexed 500 mg/m^2 every 3 weeks until disease progression or significant toxicity and continue with HAL administration given every 2 weeks (not to exceed 16 total immunizations).
  Interventions: Drug: Docetaxel; Biological: HyperAcute®-Lung Immunotherapy; Drug: Gemcitabine; Drug: Pemetrexed
- Arm 2b: HyperAcute®-Lung Immunotherapy (biweekly) (Experimental): Arm 2b: 300 Million HAL cells given by intradermal injection biweekly for 6 doses and then every month for 10 additional doses.
  Up to 16 total immunizations of 300 million immunotherapy cells until disease progression or toxicity.
  First Progression: Docetaxel 75 mg/m^2 IV given every 3 weeks or Gemcitabine 1250 mg/m^2 for 2 weeks with 1 week rest or Pemetrexed 500 mg/m^2 every 3 weeks until disease progression or significant toxicity and continue with HAL administration given every 2 weeks (not to exceed 16 total immunizations).
  Interventions: Drug: Docetaxel; Biological: HyperAcute®-Lung Immunotherapy; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: Docetaxel — Docetaxel given in Arm 1 prior to first progression on study. Given as an option of salvage therapy after first progression on study for Arms 2a and 2b.
  Other Names: Taxotere®
Biological: HyperAcute®-Lung Immunotherapy — HAL-1, HAL-2 and HAL-3 immunotherapy components.
  Up to 16 immunizations of 300 million immunotherapy cells.
  Other Names: Tergenpumatucel-L
  Arms: Arm 2a: HyperAcute®-Lung Immunotherapy (weekly); Arm 2b: HyperAcute®-Lung Immunotherapy (biweekly)
Drug: Gemcitabine — Given as an option of salvage therapy after first progression on study for Arms 1, 2a and 2b.
  Other Names: Gemzar®
Drug: Pemetrexed — Given as an option of salvage therapy after first progression on study for Arms 1, 2a and 2b.
  Other Names: Alimta®

SUMMARY:
The purpose of this study is to assess overall survival of anti-tumor immunization using HyperAcute®-Lung immunotherapy versus Docetaxel in patients with progressed or relapsed non-small cell lung cancer (NSCLC) that have been previously treated.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) remains the leading cause of cancer death in men and women in the United States. Despite advances in the treatment of advanced NSCLC in the last decade, survival outcomes remain poor. Treatment benefit from cytotoxic chemotherapy has reached a plateau and further progress will depend upon identifying novel methods to target tumor cells.

Harnessing the human immune system to target lung cancer could result in the development of effective treatment options against lung cancer and potentially enhance the effect of cytotoxic chemotherapy. Lung cancer cells produce a number of abnormal proteins or abnormal amounts of certain proteins found in normal lung cells. In some cancers, the abnormal protein expression may lead to an immune response against the cancer cells much in the way the immune system responds to an infection. In progressive lung cancer however, the immune system fails to identify or respond to these abnormalities and the cancer cells are not attacked or destroyed for reasons not yet fully understood. This clinical trial proposes a novel method to stimulate the immune system to recognize the abnormal components found in lung cancer cells and to stimulate an immune response that destroys or blocks the growth of the cancer.

This new method of treatment helps the immune system of lung cancer patients to "identify" and target the cancerous tissue. As an example, patients who receive an organ transplant to replace a damaged kidney or heart are treated with special drugs to supress their immune response from destroying or "rejecting" the transplanted organ. This "rejection" occurs when the patient's immune system responds to differences between the cells of the transplanted organ and their own immune system by attacking the foreign tissue in the same way as it would attack infected tissue. When the differences between foreign tissues and the patient's body are even larger, perhaps like differences between organs from pigs and the immune system cells of humans, the rejection is very rapid, highly destructive and the immunity it generates is long-lasting. This is called hyperacute rejection and the medicine used to immunize patients in this protocol tries to harness this response to teach a patient's immune system to fight their lung cancer just as the body would learn to reject a transplanted organ from an animal.

To do this, we have placed a mouse gene into cultured human lung cancer cell lines. These cells will express a sugar that will stimulate a strong immune response in humans. These cancer cells are irradiated to prevent any growth and then injected along with chemotherapy to patients with lung cancer. The presence of the sugar will stimulate the patient's immune system to kill the injected immunotherapy cells. As part of the process of destroying the immunotherapy cells, the patient's immune system is stimulated to identify as many differences between these cancer cells and normal human cells. This extra stimulation is thought to encourage immune responses against the lung cancer in the patient based on shared abnormalities of lung cancer immunotherapy cells and the patient's lung cancer cells.

In this experimental therapy, patients are given docetaxel or injections of an immunotherapy consisting of three types of modified lung cancer cells. We propose to test these treatments in patients with lung cancer who have progressed after initial chemotherapy to demonstrate that treatment of immunotherapy results in improved tumor stabilization or response and could potentially improve the patient's overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of non-small cell lung cancer (NSCLC). Squamous cell (epidermoid), adenocarcinoma, bronchoalveolar carcinoma, and large cell anaplastic lung carcinoma histologies are eligible as are mixed histologies of NSCLC (i.e., adenosquamous). Mixed NSCLC/small cell lung carcinoma (SCLC), and variant large and small cell lung cancer are not eligible.
* Stage IIIB (AJCC Stage IIIB - Any T,N3M0 or T4N2M0) or Metastatic (AJCC Stage IV- any T, any N, M1), progressive, recurrent or refractory NSCLC. Patients may not be eligible for other curative intent treatment (e.g., surgical resection).

For the purpose of eligibility for this trial, the above-cited disease states are defined as follows:

* Progressive NSCLC: Defined as increasing measurable disease, or the appearance of new measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria despite treatment.
* Recurrent NSCLC: Defined as the re-appearance of measurable disease, or the appearance of new measurable disease by RECIST Criteria after prior successful treatment or complete response.
* Refractory NSCLC: Defined as achieving less than a complete response and having residual measurable disease by RECIST criteria after prior treatment with chemotherapy, targeted or small molecules, monoclonal antibodies or any combination of these.
* Eastern Cooperative Oncology Group (ECOG)Performance Status ≤ 1.
* Serum albumin ≥3.0 gm/dL.
* Expected survival ≥4 months.
* Adequate organ function including:

  1. Marrow: Hemoglobin ≥10.0 dm/dL, absolute granulocyte count (AGC)≥1,000/mm^3, platelets ≥100,000/mm^3, absolute lymphocyte count ≥1000/mm^3.
  2. Hepatic: Serum total bilirubin ≤1.5 x upper limit of normal (ULN) with the exception of <2.9 mg/dL for patients with Gilbert's disease, alanine aminotransferase (ALT/SGPT) and aspartate aminotransferase (AST/SGOT) ≤2.5 x ULN.
  3. Renal: Serum creatinine (sCr) ≤1.5 x upper limit of normal, or creatinine clearance (Ccr) ≥50 mL/min.
* Measurable disease as defined by RECIST Criteria.
* Prior therapy for NSCLC that may include surgery, radiation therapy, immunotherapy and/or ≤ 2 prior chemotherapy regimens (such as neoadjuvant/adjuvant treatment), however only 1 chemotherapy regimen in the metastatic setting is allowed.
* Treatment with a single course of gefitinib(Iressa®) or erlotinib (Tarceva®), or other small molecule or targeted therapies, or monoclonal antibody therapy (excluding docetaxel) will be considered and count as prior chemotherapy.
* Patients receiving preoperative (Neoadjuvant) and postoperative adjuvant chemotherapy (within 12 weeks of surgery) with the same agent(s) will be considered to have received a single chemotherapy regimen.
* Patients must be ≥ 4 weeks since major surgery, chemotherapy (6-weeks if they were treated with a nitrosourea or mitomycin) or biotherapy/target therapies and ≥ 2 weeks since radiotherapy.
* Patients must have the ability to understand the study, its risks, side effects, potential benefits and be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* Male and female subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental drug and for one month after the last immunization.

Exclusion Criteria:

* Age < 18-years-old.
* Active central nervous system (CNS) disease, metastases or carcinomatous meningitis. Patients with CNS metastases must be at least 2 weeks status post prior therapy to the brain and be off all steroids without progressing CNS disease.
* Hypercalcemia >2.9 mmol/L, unresponsive to standard therapy (e.g., I.V. hydration, diuretics, calcitonin and/or bisphosphate therapy).
* Pregnant or nursing women due to the unknown effects of immunization on the developing fetus or newborn infant.
* Other malignancy within three years, unless the probability of recurrence is <5%. Patients curatively treated for squamous cell carcinoma and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.
* History of organ transplant, or current active immunosuppressive therapy (such as cyclosporine, tacrolimus, etc.).
* Subjects taking systemic corticosteroid therapy for any reason including replacement therapy for hypoadrenalism, are not eligible. Subjects receiving inhaled or topical corticosteroids are eligible. Decadron treatment with docetaxel is acceptable.
* Significant or uncontrolled congestive heart failure (CHF), myocardial infarction, significant ventricular arrhythmias within the last six months or significant pulmonary dysfunction.
* Active infection or antibiotics within 48 hours prior to study enrollment, including unexplained fever (temp > 38.1°C) if deemed clinically significant by the treating physician.
* Autoimmune disease (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), etc.). Patients with a remote history of asthma or mild active asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis).
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc).
* A known allergy to any component of the HyperAcute®-Lung immunotherapy or cell lines from which it is derived.
* Patients having undergone splenectomy.
* Known HIV positive.
* Subjects who received any prior treatment with docetaxel are excluded. Subjects who have received gemcitabine in first line therapy but do not have squamous cell carcinoma, will be eligible as they can receive pemetrexed for the salvage regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05-18 (Actual); Study Completion 2016-06-18 (Actual)

PRIMARY OUTCOMES:
Overall survival | Approximately 19 months, assuming a 24 month enrollment.
  The primary objective in Phase IIB and Phase III is to assess overall survival of anti-tumor immunization using HyperAcute®-Lung (HAL) Immunotherapy versus docetaxel in patients with progressed or relapsed non-small cell lung cancer (NSCLC) that have been previously treated.

SECONDARY OUTCOMES:
Dosing schedule | Approximately 19 months, assuming a 24 month enrollment.
  A secondary objective in Phase IIB is to determine the response rates of HyperAcute®-Lung (HAL) Immunotherapy given in a weekly and biweekly regimen versus docetaxel.
Tumor response rate | Approximately 19 months, assuming a 24 month enrollment.
  A secondary outcome measure in Phase IIB and Phase III is to measure tumor response including response to follow-on salvage regimens to assess chemosensitization effects.
Immunologic Response | Approximately 19 months, assuming a 24 month enrollment.
  A secondary outcome measure in Phase IIB and Phase III is to assess the immunological response of patients with lung cancer treated with HyperAcute®-Lung (HAL) Immunotherapy versus docetaxel in patients with progressed or relapsed NSCLC that have been previously treated.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Stamford Hospital, Stamford, Connecticut
  - University of Florida, Gainesville, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Cancer Center, Fairway, Kansas
  - North Mississippi Hematology and Oncology Associates at BridgePoint, Tupelo, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Richmond University Medical Center, Staten Island, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Vince Lombardi Cancer Clinic, Green Bay, Wisconsin
  - University of Wisconsin, Madison, Wisconsin